CLINICAL TRIAL: NCT07388745
Title: A Randomized Trial Comparing Erector Spinae Plane Block Versus Serratus Posterior Superior Intercostal Plane Block for Postoperative Analgesic Efficacy in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: ESPB vs SPSIP for Postoperative Analgesia After CABG
Acronym: ESP-SPSIP-CABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Merve Yaman, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSBÜ-KVC-CABG-ESPB-SPSIPB-2026
Record Dates: First submitted 2026-01-25; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Coronary Arterial Disease; Coronary Artery Bypass Grafting (CABG) Surgery; Postoperative Pain Management
Keywords: Coronary Artery Bypass Grafting; Erector Spinae Plane Block; Serratus Posterior Superior Intercostal Plane Block; Regional Anesthesia; Ultrasound-Guided Nerve Block; Postoperative Pain; Numeric Rating Scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (ESPB) (Active Comparator): Ultrasound-guided bilateral Erector Spinae Plane Block will be performed preoperatively under sedation at the T4-T5 transverse process level. A total of 20 mL of 0.25% bupivacaine will be injected per side (total 40 mL). All participants will receive standardized general anesthesia for CABG and the same postoperative multimodal analgesia protocol.
  Interventions: Procedure: Ultrasound-guided Erector Spinae Plane Block (ESPB)
- Serratus Posterior Superior Intercostal Plane Block (SPSIPB) (Experimental): Ultrasound-guided bilateral Serratus Posterior Superior Intercostal Plane Block will be performed preoperatively under sedation at the 2nd-3rd intercostal space. A total of 20 mL of 0.25% bupivacaine will be injected per side (total 40 mL). All participants will receive standardized general anesthesia for CABG and the same postoperative multimodal analgesia protocol.
  Interventions: Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block (SPSIPB)

INTERVENTIONS:
Procedure: Ultrasound-guided Erector Spinae Plane Block (ESPB) — Bilateral ultrasound-guided ESPB performed preoperatively under sedation at the T4-T5 transverse process level using 20 mL of 0.25% bupivacaine per side (total 40 mL).
  Arms: Erector Spinae Plane Block (ESPB)
Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block (SPSIPB) — Bilateral ultrasound-guided SPSIPB performed preoperatively under sedation at the 2nd-3rd intercostal space using 20 mL of 0.25% bupivacaine per side (total 40 mL).
  Arms: Serratus Posterior Superior Intercostal Plane Block (SPSIPB)

SUMMARY:
This prospective, randomized, active-controlled, double-blind, parallel-group study compares the postoperative analgesic efficacy and safety of ultrasound-guided bilateral Erector Spinae Plane Block (ESPB) versus bilateral Serratus Posterior Superior Intercostal Plane Block (SPSIPB) in adult patients (45-85 years, ASA I-III) undergoing elective coronary artery bypass graft surgery. The primary outcome is postoperative pain intensity assessed by Numeric Rating Scale (NRS) at 2, 4, 8, 16, 24, and 48 hours after surgery. Secondary outcomes include intraoperative fentanyl/remifentanil consumption, postoperative morphine consumption, patient-controlled analgesia (PCA) demand/delivery parameters (if PCA is used), need for rescue analgesics, extubation and mobilization times, peak inspiratory flow measured by incentive spirometry at predefined time points, ICU and hospital length of stay, recovery quality (QoR-15 at 0, 24, and 48 hours), mortality, and block-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-85 years
* Scheduled for elective coronary artery bypass graft (CABG) surgery
* American Society of Anesthesiologists (ASA) I-II-III
* Patients who provide written informed consent and agree to participate in the study

Exclusion Criteria:

* Emergency cases
* ASA IV-V
* Known allergy to local anesthetics
* Coagulopathy (platelet count <100,000/mm³, INR >1.5, aPTT >1.5× normal)
* Infection at the block injection site
* Pregnancy
* Patients who do not provide written informed consent or decline to participate after being informed

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | 2, 4, 8, 16, 24, and 48 hours after surgery
  Pain intensity will be assessed using the Numerical Rating Scale (NRS), ranging from 0 to 10, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Cumulative postoperative opioid consumption | First 24 hours after surgery
  Total opioid dose for analgesia converted to IV morphine equivalents.
Need for rescue analgesia | Up to 48 hours after surgery
  Proportion of participants requiring rescue analgesics in addition to the standardized protocol.
Quality of Recovery (QoR-15) score | Baseline (preoperative), postoperative 24 hours, and 48 hours after surgery
  "The Quality of Recovery-15 questionnaire (QoR-15) is a patient-reported measure consisting of 15 items. Each item is scored from 0 (unfavourable) to 10 (favourable), resulting in a total score ranging from 0 to 150. Higher total scores indicate better postoperative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yaman, Assistant Professor, Principal Investigator — Kütahya Health Sciences University

IPD SHARING:
Plan to Share IPD: No